CLINICAL TRIAL: NCT00626470
Title: A Prospective Randomised Study of Unstable Trochanteric Femur Fractures Treated With Dynamic Hip Screw With and Without a Trochanter Support Plate
Brief Title: Prospective Trial on Trochanteric Femur Fractures Treated With or Without a Trochanter Support Plate
Acronym: TSP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSP Study
Record Dates: First submitted 2008-02-15; First posted 2008-02-29 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Femoral Fractures
Keywords: Trochanter; Femur; Fracture
MeSH Terms: conditions — Femoral Fractures; Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- -TSP (Active Comparator): Patients operated without TSP
  Interventions: Procedure: Addition of TSP to DHS
- +TSP (Active Comparator): Patients operated with TSP
  Interventions: Procedure: Addition of TSP to DHS

INTERVENTIONS:
Procedure: Addition of TSP to DHS — All patients operated with DHS. Of these two groups. One operated with TSP and one without.

SUMMARY:
Fractures just below the hip often are treated with a so called Gliding Screw and Plate (DHS). Recently a new additional plate called a Trochanter Support Plate (TSP) which attaches to the DHS has become available which is claimed to give extra support to the fracture. In a prospective randomised study we wish to test the hypothesis that the TSP does not give any additional stability to the fracture treated with the DHS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unstable trochanteric femur fracture.(Evans-Jensen class.3-5)
* (can include; Patients with cognitive problems (ie. dementia etc)

Exclusion Criteria:

* Patients with pathological fractures
* Multitrauma patients
* Patients not able to walk before the fracture
* Under 19 years old.
* Patients with fractures needing other treatments than gliding hip screws
* Reverse oblique fractures.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Fracture movement postoperatively | One year

SECONDARY OUTCOMES:
Reoperation | One year
Pain postoperatively | one year
Hip function postoperatively | one year
Fracture healing | one year
complications postoperatively | one year

CONTACTS AND LOCATIONS:
Overall Officials: James Haddon, MD, Principal Investigator — St. Olavs Hospital
Locations (1):
- Ortopaedic Department, St.Olavs Hospital, Trondheim, Norway